CLINICAL TRIAL: NCT00521560
Title: Phase I/II Study Concomitant High-Dose Radio-Immuno- and Chemotherapy With Simultaneous Application of Zevalin and BEAM Followed by Autologous Peripheral Stem Cell Transplantation in Relapsed and Refractory CD 20+ Non-Hodgkin's Lymphoma
Brief Title: A Study of Zevalin and Simultaneous Application of BEAM High-dose Chemotherapy Followed by Autologous Stem Cell Transplantation in Refractory and Relapsed Aggressive Non-Hodgkin Lymphomas
Acronym: escZ-BEAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2004-R4; DSHNHL 2004-R4
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Primary Non-Hodgkin-Lymphoma; Refractory Non-Hodgkin-Lymphoma; CD20+ Aggressive Non-Hodgkin's Lymphoma
Keywords: High-Dose Radio-Immuno- and Chemotherapy; stem cell transplantation; 90Y-Ibritumomab-Tiuxetan
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Zevalin

INTERVENTIONS:
Drug: Zevalin — All applications of 90Y-Ibritumomab-Tiuxetan will be preceded by rituximab infusions at a dose of 250 mg/m2 at days -21 and day -14 (DL1) or day -12 (DL2) or day -10 (DL3-5), respectively.
  High dose therapy will be given as BEAM
  Other Names: 90Y-Ibritumomab-Tiuxetan

SUMMARY:
Phase II Study Concomitant High-Dose Radio-Immuno- and Chemotherapy with simultaneous application of Zevalin and BEAM followed by autologous peripheral stem cell transplantation in relapsed and refractory CD 20+ Non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years
* Risk group: 1) Progression on primary therapy 2) Initial or subsequent relapse
* Histology: Diagnosis of relapsed aggressive non-Hodgkin lymphoma, whenever possible confirmed by an excision biopsy of a lymph node or by a sufficiently large biopsy of an extranodal site if no lymph node lesion is present. The expression of the CD20 antigen must be demonstrated in the primary lesion or in the relapse. Specifically, the following entities can be treated in this study:

B-NHL:

Grade III B follicular lymphoma Diffuse B-cell lymphoma centroblastic immunoblastic plasmoblastic anaplastic-large-cell T-cell rich B-cell lymphoma Primary effusion lymphoma Intravascular B-cell lymphoma Primary mediastinal B-cell lymphoma Mantle cell lymphoma, blastoid Variants of Burkitt's lymphoma Aggressive marginal zone lymphoma (monocytoid)

* General condition: General condition ECOG 0-3 (Karnofsky: 40 - 100 %); for definition see Annex 14.10
* Presence of declaration of participation of the center and the patient's written consent form

Exclusion Criteria:

* Prior mediastinal or extensive abdominal irradiation
* Prior high-dose therapy and autologous stem cell transplantation
* Impairment of renal function (creatinine > 2.5 mg/dL, creatinine clearance < 20 mL/min)
* Impairment of hepatic function (bilirubin > 2.0 mg/dL, cholinesterase [CHE] < 2000 U/L)
* Impairment of pulmonary function (transfer lung factor for CO [TLCO] < 50 %, forced expiratory volume in 1 sec [FEV1] < 60 %, vital capacity [VC] < 60 %)
* Relevant deterioration of the above organ functions on salvage therapy
* Failure of stem cell mobilization
* Active viral hepatitis
* HIV infection
* Other active or not conclusively curatively treated malignoma
* Severe concomitant psychiatric illness or suspected lack of patient compliance
* Pregnancy or unreliable contraception
* Highly dynamic progress of lymphoma (lactate dehydrogenase [LDH] > 1.5 x upper limit of normal [ULN]) after salvage therapy immediately prior to radioimmunotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-03; Primary Completion 2009-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the highest achievable dose level of 90Y-Zevalin administered immediately before BEAM high-dose therapy and followed by autologous stem cell transplantation. | 3 Year

SECONDARY OUTCOMES:
Treatment related mortality (TRM), freedom from progression (FFP), Survival (OS), progression free survival (PFS) grade III -IV toxicity (CTC) on lung, liver and kidney | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Glass, Prof. Dr., Study Director — German Society of Cancer e.V.; Martin Gramatzki, MD PhD, Principal Investigator — Städtisches Krankenhaus Kiel, II. Med. Uniklinik, Kiel, Germany; Mattias Witzens Harig, MD PhD, Principal Investigator — Abteilung Innere Medizin V, Hämatologie, Onkologie, Heidelberg, Germany; Bernd Hertenstein, MD PhD, Principal Investigator — Klinikum Bremen-Mitte gGmbH, Medizinische Klinik I, Bremen, Germany; Georg Heß, MD PhD, Principal Investigator — III Med., Schwerpunkt Hämatologie / Onkologie, Mainz, Germany; Dorothea Kofahl-Krause, MD PhD, Principal Investigator — MHH, Hämatologie, Hämostaseologie und Onkologie, Hannover, Germany; Norbert Schmitz, MD PhD, Principal Investigator — Asklepios Klinik St. Georg, Hämatologische Abt., Hamburg, Germany; Jörg Schubert, MD PhD, Principal Investigator — Universitätskliniken d. Saarlandes, Med. I, Homburg/Saar, Germany; Lutz Uharek Uharek, MD PhD, Principal Investigator — Charité - Campus Benjamin Franklin, Med. III, Berlin, Germany
Locations (1):
- Institut für anwendungsorientierte Forschung und klinische Studien (IFS GmbH), Göttingen, Germany